CLINICAL TRIAL: NCT05678998
Title: A Phase 1 (First-In-Human [FIH]), Multi-Site, Dose Escalation and Expansion Study of WTX-330 in Adult Patients With Advanced or Metastatic Solid Tumors or Lymphoma
Brief Title: WTX-330 in Patients With Advanced or Metastatic Solid Tumors or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Werewolf Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WTX-330x2101
Record Dates: First submitted 2022-12-09; First posted 2023-01-10 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Advanced or Metastatic Solid Tumors; Non-Hodgkin Lymphoma
Keywords: WTX-330; Cancer; Immunotherapy; Interleukin-12; IL-12; Checkpoint inhibitor resistance
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- WTX-330 dose escalation (Experimental): Patients with relapsed/refractory advanced or metastatic solid tumors
  Interventions: Drug: WTX-330
- WTX-330 dose expansion in patients for whom CPI therapy is indicated (Arm A) (Experimental): WTX-330 dose expansion in patients with tumor types for which a CPI is indicated/approved who demonstrate primary or secondary resistance to an anti-PD(L)1-based regimen
  Interventions: Drug: WTX-330
- WTX-330 dose expansion in patients for whom CPI therapy is not indicated (Arm B) (Experimental): WTX-330 dose expansion in patients with tumor types for which a CPI is not indicated/ approved
  Interventions: Drug: WTX-330

INTERVENTIONS:
Drug: WTX-330 — Investigation Product

SUMMARY:
A first-in-human, Phase 1, open-label, multicenter study of WTX-330 administered as a monotherapy to patients with advanced or metastatic solid tumors or non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, open-label, multicenter study to evaluate the safety, tolerability and preliminary efficacy of WTX-330, a conditionally-activated IL-12 prodrug, when administered as a monotherapy to patients with advanced or metastatic solid tumors or non-Hodgkin lymphoma. Dose escalation will be conducted in patients with advanced and/or metastatic solid tumors who are refractory to all standard of care therapies. Dose expansion will be conducted in two arms: Arm A will enroll patients with indications for which a checkpoint inhibitor (CPI) is indicated/approved who demonstrate primary or secondary resistance to an anti-PD(L)1 treatment regimen, and Arm B will enroll patients with tumor types for which CPI therapy is not indicated/approved.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Dose Escalation: A diagnosis of a relapsed/refractory advanced or metastatic solid tumor for which the patient has progressed on or is intolerant of standard therapy, or for whom no standard therapy with proven benefit exists.
3. Dose Expansion: A diagnosis of a relapsed/refractory advanced or metastatic malignancy for which the patient has progressed on or is intolerant of standard therapy, or for whom no standard therapy with proven benefit exists. For Arm A, patients must have a tumor type for which a CPI is indicated/approved and demonstrate primary or secondary resistance to a standard of care anti-PD(L)1-based treatment regimen. For Arm B, patients must have a solid tumor type for which a CPI is not indicated/approved or non-Hodgkin lymphoma.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. At least one measurable lesion per RECIST 1.1 or an evaluable lesion per Lugano classification (for lymphoma).
6. Agrees to undergo a pre-treatment and on-treatment biopsy of a primary or metastatic solid tumor or lymphoma lesion.
7. HIV-infected patients must be on antiretroviral therapy and have well-controlled disease.
8. Adequate organ and bone marrow function.
9. Willingness of men and women of reproductive potential to use highly effective birth control for the duration of treatment and for 4 months following the last dose of study drug.
10. Additional criteria may apply.

Exclusion Criteria:

1. A history of another active malignancy (i.e., a second cancer) within the previous 2 years, except for localized cancers that are not related to the current cancer being treated, are considered cured, and, in the opinion of the Investigator, present a low risk of recurrence. These exceptions include but are not limited to basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
2. Received prior treatment with IL-12, including by intratumoral injection.
3. Patients with primary CNS malignancies.
4. Presence of CNS metastases that are symptomatic and/or require local CNS directed therapy (such as XRT or surgery) or increasing doses of corticosteroids within 2 weeks prior to the first dose of study drug. Patients with treated brain metastases should be neurologically stable and receiving ≤ 10 mg per day of prednisone or equivalent prior to study entry.
5. Significant cardiovascular disease.
6. Significant electrocardiogram (ECG) abnormalities
7. Active autoimmune disease requiring systemic treatment in the past 2 years.
8. Diagnosis of immunodeficiency, on immunosuppressive therapy, or receiving chronic systemic or enteric steroid therapy (dose > 10 mg/day of prednisone or equivalent).
9. Prior receipt of an allogeneic stem cell transplant or allogeneic CAR-T cell therapy.
10. Major surgery (excluding placement of vascular access) within 2 weeks prior to the first dose of study drug.
11. Investigational agent or anticancer therapy (including chemotherapy, biologic therapy, immunotherapy, anticancer Chinese medicine, or anticancer herbal remedy) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug.
12. Radiotherapy within 2 weeks of the start of study treatment. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
13. Any unresolved toxicities from prior therapy greater than NCI-CTCAE version 5.0 Grade 1 at the time of starting study drug with the exception of alopecia and Grade 2 platinum therapy-related neuropathy.
14. Use of sensitive substrates of major CYP450 isozymes.
15. Any illness, medical condition, organ system dysfunction, or social situation (including mental illness or substance abuse), that may interfere with a patient's ability to sign the ICF, adversely affect the patient's ability to cooperate and participate in the study, or compromise interpretation of study results.
16. Received a live vaccine within 30 days of the first dose of study drug.
17. Active, uncontrolled systemic bacterial, viral, or fungal infection.
18. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
19. Active infection with hepatitis B as determined by hepatitis B surface antigen and hepatitis B core antibody, or hepatitis B virus deoxyribonucleic acid (DNA) by quantitative polymerase chain reaction (qPCR) testing.
20. Active infection with hepatitis C as determined by hepatitis C virus (HCV) antibody or HCV RNA by qPCR testing.
21. Pregnant or lactating.
22. History of hypersensitivity to any of the study drug components.
23. Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - HonorHealth, Scottsdale, Arizona
  - Emory Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Mass General Hospital, Boston, Massachusetts
  - Facility Name: Roswell Park Comprehensive Cancer Care, Buffalo, New York
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - NEXT Oncology, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on their oncological history at 9 clinical research sites in the United States.
Pre-assignment Details: 36 potential participants underwent screening, 11 were screened out, and 25 were included in the trial.
Groups:
- WTX-330 Dose Escalation - 0.016 mg/kg: Patients with relapsed/refractory advanced or metastatic solid tumors received a dose of 0.016 mg/kg on Days 1 and 15 (i.e., every 2 weeks, Q2W) of 28-day treatment cycle
- WTX-330 Dose Escalation - 0.024 mg/kg: Patients with relapsed/refractory advanced or metastatic solid tumors received a dose of 0.024 mg/kg on Days 1 and 15 (i.e., every 2 weeks, Q2W) of 28-day treatment cycle
- WTX-330 Dose Escalation - 0.032 mg/kg: Patients with relapsed/refractory advanced or metastatic solid tumors received a dose of 0.032 mg/kg on Days 1 and 15 (i.e., every 2 weeks, Q2W) of 28-day treatment cycle
- WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg: WTX-330 dose expansion in patients with tumor types for which a CPI is indicated/approved who demonstrate primary or secondary resistance to an anti-PD(L)1-based regimen. Expansion Dose was 0.024 mg/kg.
- WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg: WTX-330 dose expansion in patients with tumor types for which a CPI is not indicated/ approved. Expansion Dose was 0.024 mg/kg.
Period: Overall Study
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg
Started | 3 | 3 | 5 | 5 | 9
Completed | 2 | 2 | 2 | 0 | 2
Not Completed | 1 | 1 | 3 | 5 | 7
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 3 | 4
Not completed — Other | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg: WTX-330 dose expansion in patients with tumor types for which a CPI is indicated/approved who demonstrate primary or secondary resistance to an anti-PD(L)1-based regimen
- WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg: WTX-330 dose expansion in patients with tumor types for which a CPI is not indicated/ approved
- Total: Total of all reporting groups
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | Total
Number analyzed (Participants) | 3 | 5 | 9 | 3 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.26) | 60.6 (11.55) | 68.2 (7.90) | 65.00 (11.00) | 61.8 (10.13) | 64.4 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 2 | 1 | 12
  Male | 1 | 3 | 4 | 1 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2
  White | 1 | 5 | 8 | 3 | 4 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 1 | 5 | 9 | 2 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle of treatment with WTX-330 and meets any of the criteria included in the protocol
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 0 | 1

2. Primary Outcome: Incidence of Treatment Emergent Adverse Events
Description: AEs were graded and documented in accordance with NCI-CTCAE version 5.0
Time Frame: 24 months
Population: Safety Analysis Set included all participants
Measure: Count of Participants; unit: Participants
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A) | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 9
Participants
  TEAE | 3 | 3 | 5 | 5 | 9
  TEAEs Related to WTX-330 | 3 | 3 | 5 | 5 | 9
  Grade 3 or Higher TEAEs | 1 | 3 | 4 | 4 | 8
  Grade 3 or Higher TEAEs Related to WTX-330 | 1 | 2 | 4 | 3 | 5
  Serious TEAEs | 0 | 1 | 2 | 3 | 8
  Serious TEAEs Related to WTX-330 | 0 | 1 | 1 | 1 | 5

3. Primary Outcome: Incidence of Changes in Clinical Laboratory Abnormalities
Description: Change from baseline is provided as baseline grade or "normal/low/high" and worst post-baseline grade.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A) | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B)
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 9
Participants
  Anemia: Grade 0 - Grade 0 | 0 | 0 | 0 | 1 | 0
  Anemia: Grade 0 - Grade 1 | 0 | 0 | 3 | 0 | 0
  Anemia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 1
  Anemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 1 - Grade 1 | 2 | 0 | 1 | 1 | 3
  Anemia: Grade 1 - Grade 2 | 1 | 2 | 0 | 0 | 4
  Anemia: Grade 1 - Grade 3 | 0 | 1 | 0 | 1 | 0
  Anemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 2 - Grade 2 | 0 | 0 | 1 | 1 | 1
  Anemia: Grade 2 - Grade 3 | 0 | 0 | 0 | 1 | 0
  Anemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Anemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Anemia: Missing | 0 | 0 | 0 | 0 | 0
  Anemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Anemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Anemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Anemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Anemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Anemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Anemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 - Grade 0 | 1 | 0 | 2 | 2 | 0
  Hypoalbuminemia: Grade 0 - Grade 1 | 2 | 2 | 2 | 0 | 6
  Hypoalbuminemia: Grade 0 - Grade 2 | 0 | 1 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 - Grade 2 | 0 | 0 | 1 | 1 | 3
  Hypoalbuminemia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 - Grade 2 | 0 | 0 | 0 | 2 | 0
  Hypoalbuminemia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Missing | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 0 - Grade 0 | 3 | 2 | 5 | 5 | 8
  Hypoglycemia: Grade 0 - Grade 1 | 0 | 1 | 0 | 0 | 0
  Hypoglycemia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 1
  Hypoglycemia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Missing | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 0 - Grade 0 | 2 | 1 | 1 | 1 | 6
  Hypokalemia: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 0 - Grade 2 | 0 | 1 | 4 | 4 | 2
  Hypokalemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 - Grade 2 | 1 | 0 | 0 | 0 | 1
  Hypokalemia: Grade 2 - Grade 3 | 0 | 1 | 0 | 0 | 0
  Hypokalemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Missing | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 0 - Grade 0 | 1 | 2 | 3 | 4 | 7
  Hypomagnesemia: Grade 0 - Grade 1 | 1 | 0 | 1 | 0 | 2
  Hypomagnesemia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 - Grade 1 | 1 | 1 | 1 | 1 | 0
  Hypomagnesemia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Missing | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 0 - Grade 0 | 2 | 0 | 1 | 1 | 2
  Hyponatremia: Grade 0 - Grade 1 | 0 | 2 | 3 | 1 | 1
  Hyponatremia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 0 - Grade 3 | 0 | 1 | 0 | 2 | 3
  Hyponatremia: Grade 1 - Grade 0 | 1 | 0 | 0 | 0 | 1
  Hyponatremia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 1
  Hyponatremia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 1 - Grade 3 | 0 | 0 | 1 | 0 | 1
  Hyponatremia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 4 - Grade 1 | 0 | 0 | 0 | 1 | 0
  Hyponatremia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Missing | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 0 - Grade 0 | 0 | 1 | 1 | 3 | 1
  Lymphocyte count decreased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased: Grade 0 - Grade 2 | 0 | 0 | 1 | 1 | 0
  Lymphocyte count decreased: Grade 0 - Grade 3 | 2 | 1 | 3 | 0 | 1
  Lymphocyte count decreased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 - Grade 3 | 0 | 1 | 0 | 0 | 3
  Lymphocyte count decreased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 - Grade 3 | 1 | 0 | 0 | 1 | 1
  Lymphocyte count decreased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 2
  Lymphocyte count decreased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Missing | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 0 - Grade 0 | 1 | 1 | 2 | 2 | 4
  Platelet count decreased: Grade 0 - Grade 1 | 1 | 2 | 2 | 3 | 2
  Platelet count decreased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 2
  Platelet count decreased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 1 - Grade 2 | 1 | 0 | 1 | 0 | 1
  Platelet count decreased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Missing | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 0 - Grade 0 | 0 | 1 | 1 | 3 | 3
  White blood cell decreased: Grade 0 - Grade 1 | 0 | 0 | 0 | 1 | 0
  White blood cell decreased: Grade 0 - Grade 2 | 2 | 1 | 2 | 0 | 3
  White blood cell decreased: Grade 0 - Grade 3 | 1 | 1 | 2 | 1 | 1
  White blood cell decreased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 1
  White blood cell decreased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 1
  White blood cell decreased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Missing | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 0 - Grade 0 | 1 | 1 | 2 | 1 | 5
  Activated partial thromboplastin time prolonged: Grade 0 - Grade 1 | 1 | 1 | 1 | 2 | 0
  Activated partial thromboplastin time prolonged: Grade 0 - Grade 2 | 1 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 0 - Grade 3 | 0 | 0 | 1 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 1 - Grade 1 | 0 | 1 | 0 | 0 | 2
  Activated partial thromboplastin time prolonged: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 1
  Activated partial thromboplastin time prolonged: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 2 - Grade 3 | 0 | 0 | 0 | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Missing | 0 | 0 | 1 | 1 | 1
  Activated partial thromboplastin time prolonged: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 0 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Missing | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Low - Grade 0 | 0 | 0 | 0 | 1 | 0
  Alanine aminotransferase increased: Normal - Grade 0 | 0 | 2 | 1 | 1 | 3
  Alanine aminotransferase increased: Normal - Grade 1 | 3 | 1 | 3 | 1 | 4
  Alanine aminotransferase increased: Normal - Grade 2 | 0 | 0 | 0 | 2 | 1
  Alanine aminotransferase increased: Normal - Grade 3 | 0 | 0 | 1 | 0 | 0
  Alanine aminotransferase increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: High - Grade 1 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 0 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Missing | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Normal - Grade 0 | 0 | 2 | 0 | 1 | 2
  Alkaline phosphatase increased: Normal - Grade 1 | 0 | 0 | 3 | 0 | 1
  Alkaline phosphatase increased: Normal - Grade 2 | 0 | 0 | 1 | 1 | 0
  Alkaline phosphatase increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: High - Grade 0 | 3 | 0 | 1 | 2 | 4
  Alkaline phosphatase increased: High - Grade 1 | 0 | 0 | 0 | 0 | 2
  Alkaline phosphatase increased: High - Grade 2 | 0 | 1 | 0 | 1 | 0
  Alkaline phosphatase increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Missing | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: Low - Grade 0 | 0 | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased: Normal - Grade 0 | 0 | 1 | 0 | 0 | 1
  Aspartate aminotransferase increased: Normal - Grade 1 | 1 | 2 | 3 | 2 | 4
  Aspartate aminotransferase increased: Normal - Grade 2 | 0 | 0 | 0 | 1 | 1
  Aspartate aminotransferase increased: Normal - Grade 3 | 0 | 0 | 1 | 1 | 0
  Aspartate aminotransferase increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: High - Grade 1 | 2 | 0 | 0 | 1 | 2
  Aspartate aminotransferase increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: High - Grade 3 | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased: Grade 0 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Missing | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: Normal - Grade 0 | 1 | 1 | 2 | 2 | 5
  Blood bilirubin increased: Normal - Grade 1 | 2 | 1 | 2 | 3 | 1
  Blood bilirubin increased: Normal - Grade 2 | 0 | 1 | 1 | 0 | 1
  Blood bilirubin increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: High - Grade 1 | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 0 - Grade 0 | 2 | 2 | 4 | 4 | 5
  Creatinine increased: Grade 0 - Grade 1 | 1 | 0 | 0 | 1 | 0
  Creatinine increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 2
  Creatinine increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 1 - Grade 1 | 0 | 1 | 1 | 0 | 1
  Creatinine increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 1
  Creatinine increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Missing | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Creatinine increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 0 - Grade 0 | 2 | 1 | 1 | 1 | 6
  GGT increased: Grade 0 - Grade 1 | 1 | 1 | 3 | 2 | 2
  GGT increased: Grade 0 - Grade 2 | 0 | 0 | 1 | 1 | 1
  GGT increased: Grade 0 - Grade 3 | 0 | 1 | 0 | 1 | 0
  GGT increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  GGT increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  GGT increased: Missing | 0 | 0 | 0 | 0 | 0
  GGT increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  GGT increased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  GGT increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  GGT increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  GGT increased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  GGT increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  GGT increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 - Grade 0 | 3 | 3 | 5 | 5 | 9
  Hemoglobin increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Missing | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 0 - Grade 0 | 3 | 3 | 5 | 5 | 8
  Hyperkalemia: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 1
  Hyperkalemia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Missing | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 0 - Grade 0 | 3 | 3 | 4 | 5 | 9
  Hypermagnesemia: Grade 0 - Grade 1 | 0 | 0 | 1 | 0 | 0
  Hypermagnesemia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Missing | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 0 - Grade 0 | 2 | 3 | 5 | 5 | 9
  Hypernatremia: Grade 0 - Grade 1 | 1 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Missing | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 0 - Grade 0 | 2 | 1 | 3 | 3 | 2
  INR increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 3
  INR increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 0 - Grade 3 | 0 | 1 | 0 | 0 | 0
  INR increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 2 | 1
  INR increased: Grade 1 - Grade 2 | 0 | 0 | 1 | 0 | 2
  INR increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 2 - Grade 2 | 1 | 1 | 1 | 0 | 1
  INR increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  INR increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  INR increased: Missing | 0 | 0 | 0 | 0 | 0
  INR increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  INR increased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  INR increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  INR increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  INR increased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  INR increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  INR increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 - Grade 0 | 3 | 3 | 5 | 5 | 9
  Lymphocyte count increased: Grade 0 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 1 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 1 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 1 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 1 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 1 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 - Grade 4 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Missing | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Low - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Normal - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Normal - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Normal - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Normal - Grade 3 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: High - Grade 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: High - Grade 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: High - Grade 2 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: High - Grade 3 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Investigator-assessed Objective Response Rate (ORR) by RECIST 1.1 and Immune ORR by iRECIST (for Solid Tumors) or Response by Lugano Criteria (for Lymphomas)
Description: RECIST = Response Evaluation Criteria in Solid Tumors
Time Frame: 24 months
Population: The overall number of participants analyzed is lower than the overall study population, as the efficacy evaluable analysis set does not include all enrolled participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 7
Percent of participants
  ORR by RECIST | 0 [0 to 70.8] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 0 [0 to 52.2] | 0 [0 to 41.0]
  immune ORR by iRECIST | 0 [0 to 70.8] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 0 [0 to 52.2] | 0 [0 to 41.0]

5. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 1 - C Max
Description: PK described by maximum concentration. Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Population: Comprehensive PK was only assessed for the dose-escalation arms. Therefore, only the 3 dose-escalation arms are represented in these analyses, and not the two expansion arms.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
mcg/ml | 0.2773 (0.11684) | 0.4290 (0.29465) | 0.8624 (0.17688)

6. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 1 - Time of Maximum Concentration Observation
Description: PK described by time to maximum concentration. Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
h | 2.40 (3.637) | 2.93 (4.561) | 3.26 (1.668)

7. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 1 - Half Life
Description: PK described by Half-Life Lambda z. Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: day
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day | 2.1886 (1.23394) | 2.7083 (1.00754) | 3.3463 (1.48342)

8. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 1 - AUC
Description: PK described by Area Under Curve (0-14 day). Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose.
Time Frame: 14 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: day*mcg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day*mcg/ml | 0.7585 (0.50363) | 1.1952 (0.84243) | 1.7270 (0.75076)

9. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 2 - C Max
Description: PK described by maximum concentration. Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Population: Comprehensive PK was only assessed for the dose-escalation arms. Therefore, only the 3 dose-escalation arms are represented in these analyses, and not the two expansion arms.
  Overall Number of Participants Analyzed is lower for cycle 2, as not all participants continued on study and not all samples were available.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
mcg/ml | 0.3210 (0.04950) | 0.6272 (0.60613) | 1.0748 (0.70201)

10. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 2 - Time of Maximum Concentration Observation
Description: PK described by time to maximum concentration. Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
h | 0.30 (0) | 1.40 (1.992) | 2.15 (2.136)

11. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 2 - Half Life
Description: PK described by Half-Life Lambda z. Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
day | 3.3296 (0.34454) | 2.8809 (1.73910) | 4.0216 (1.06686)

12. Secondary Outcome: Plasma Concentrations of WTX-330 Cycle 2 - AUC
Description: PK described by Area Under Curve (0-14 day). Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose.
Time Frame: 14 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*mcg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
day*mcg/ml | 1.0247 (0.14275) | 0.8744 (0.51499) | 1.8042 (0.80145)

13. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 1 - C Max
Description: as for outcome 5
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
pg/ml | 1434.7 (694.10) | 2298.0 (1434.71) | 3022.0 (787.48)

14. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 1 - Time of Maximum Concentration Observation
Description: as for outcome 6
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
h | 4.90 (1.473) | 5.23 (2.065) | 6.48 (2.182)

15. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 1 - Half Life
Description: as for outcome 7
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: day
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day | 3.2138 (1.33405) | 3.2643 (1.26642) | 2.4809 (0.75436)

16. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 1 - AUC
Description: PK described by Area Under Curve (0-14 day). Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose.
Time Frame: 14 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: day*pg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 3 | 3 | 5
day*pg/ml | 3221.5 (1879.29) | 5144.7 (3395.29) | 5986.4 (2336.59)

17. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 2 - C Max
Description: as for outcome 9
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
pg/ml | 1331.5 (26.16) | 2165.7 (1933.23) | 3292.8 (2236.70)

18. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 2 - Time of Maximum Concentration Observation
Description: as for outcome 10
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
h | 13.80 (13.435) | 0.27 (0.058) | 2.95 (1.782)

19. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 2 - Half Life
Description: as for outcome 11
Time Frame: 0, 4, 8, 24, 48, and 168 hours post-dose on Day 1 of Cycle 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
day | 2.2540 (0.92905) | 3.8541 (0.92348) | 2.7120 (1.54085)

20. Secondary Outcome: Plasma Concentrations of IL-12 Cycle 2 - AUC
Description: PK described by Area Under Curve (0-14 day). Sample collection timepoints: 0, 4, 8, 24, 48, and 168 hours post-dose.
Time Frame: 14 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*pg/ml
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg
Number analyzed (Participants) | 2 | 3 | 4
day*pg/ml | 3569.4 (636.45) | 1957.5 (635.67) | 4349.9 (1530.39)

21. Secondary Outcome: Antidrug Antibody (ADA) Occurrence
Description: ADA were measured at Baseline and Post Baseline. "Positive" post baseline applies if at least one post-baseline value was positive.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 9
Participants
  ADA at Baseline: Negative | 2 | 3 | 4 | 5 | 8
  ADA at Baseline: Positive | 1 | 0 | 1 | 0 | 1
  ADA at Baseline: Unknown | 0 | 0 | 0 | 0 | 0
  ADA post Baseline: Negative | 2 | 2 | 2 | 3 | 5
  ADA post Baseline: Positive | 1 | 1 | 2 | 0 | 0
  ADA post Baseline: Unknown | 0 | 0 | 1 | 2 | 4

ADVERSE EVENTS:
Time Frame: AEs were collected from the signing of the ICF for a median duration of 86 days (min 37, max 219)
Description: All AEs were graded and documented in accordance with NCI-CTCAE version 5.0
Arm/Group | WTX-330 Dose Escalation - 0.016 mg/kg | WTX-330 Dose Escalation - 0.024 mg/kg | WTX-330 Dose Escalation - 0.032 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 3/5 | 5/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/5 | 3/5 | 8/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WTX-330 Dose Escalation - 0.016 mg/kg (N=3) | WTX-330 Dose Escalation - 0.024 mg/kg (N=3) | WTX-330 Dose Escalation - 0.032 mg/kg (N=5) | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg (N=5) | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg (N=9)
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 1 | 0 | 4
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Malignant melanoma of sites other than skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WTX-330 Dose Escalation - 0.016 mg/kg (N=3) | WTX-330 Dose Escalation - 0.024 mg/kg (N=3) | WTX-330 Dose Escalation - 0.032 mg/kg (N=5) | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Indicated (Arm A); 0.024 mg/kg (N=5) | WTX-330 Dose Expansion in Patients for Whom CPI Therapy is Not Indicated (Arm B); 0.024 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 5 | 0 | 3
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 1 | 0 | 4 | 2 | 6
Fatigue (General disorders) | 2 | 2 | 3 | 1 | 3
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 3 | 3 | 4
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 2 | 2 | 3 | 2
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 3 | 1 | 4
Ammonia increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 3 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cortisol decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 3 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Malignant melanoma of sites other than skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT05678998/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT05678998/SAP_001.pdf